CLINICAL TRIAL: NCT05809622
Title: Comparison of the Effectiveness of Upper Extremity-based Exercises and Elbow-focused Exercises in Lateral Elbow TendiNopathy
Brief Title: Upper Extremity-based Exercises and Elbow-focused Exercises in LET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Pelin Tiryaki, Physical Therapist, MSc, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-05
Record Dates: First submitted 2022-06-06; First posted 2023-04-12 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Lateral Epicondylitis; Elbow Tendinopathy
Keywords: tendinopathy; elbow
MeSH Terms: conditions — Tennis Elbow; Elbow Tendinopathy; Tendinopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shoulder and scapular strengthening group (Experimental)
  Interventions: Behavioral: Scapular and rotator cuff muscles strengthening
- Control group (Active Comparator)
  Interventions: Behavioral: Elbow focused rehabilitation

INTERVENTIONS:
Behavioral: Elbow focused rehabilitation — * Patient education
  * Activity modification
  * 2 days/week, 8 weeks in total
  * Exercises for the wrist extensor tendon, especially the extensor carpi radialis brevis (EKRB) (stretching + strengthening)
  Arms: Control group
Behavioral: Scapular and rotator cuff muscles strengthening — * Patient education
  * Activity modification
  * 2 days/week, 8 weeks in total
  * Exercises for the wrist extensor tendon, especially the extensor carpi radialis brevis (EKRB) (stretching + strengthening)
  * Scapular stabilizer muscle + rotator cuff (RM) strengthening
  Arms: Shoulder and scapular strengthening group

SUMMARY:
The aim of the study is to investigate the effects of rotator cuff and scapular muscle strengthening exercises applied in addition to the 8-week elbow focused rehabilitation program in lateral elbow tendinopathy, by comparing it with the elbow focused rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Cases are between the ages of 18-65
* Getting a diagnosis of unilateral lateral elbow tendinopathy
* At least two positive Thomsen, Maudsley's Mill's and Cozen tests on clinical examination
* Continuing symptoms for at least 3 months
* The absence of any chronic disease that would prevent participation in the treatment program

Exclusion Criteria:

* History of trauma or surgery in the involved elbow joint
* Having orthopedic problems in the cervical spine, shoulder joint or wrist
* To have participated in the rehabilitation program in the last 3 months
* Corticosteroid injection application in the last 3 months
* Systemic arthritis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient-Rated Tennis Elbow Evaluation (PRTEE) | Baseline
  The Patient-Rated Tennis Elbow Evaluation questionnaire (PRTEE) is a specific questionnaire available for assessing the health status of patients with lateral epicondylitis.
Patient-Rated Tennis Elbow Evaluation (PRTEE) | 8th week
  The Patient-Rated Tennis Elbow Evaluation questionnaire (PRTEE) is a specific questionnaire available for assessing the health status of patients with lateral epicondylitis.
Patient-Rated Tennis Elbow Evaluation (PRTEE) | 16th week
  The Patient-Rated Tennis Elbow Evaluation questionnaire (PRTEE) is a specific questionnaire available for assessing the health status of patients with lateral epicondylitis.
Patient-Rated Tennis Elbow Evaluation (PRTEE) | 6th month
  The Patient-Rated Tennis Elbow Evaluation questionnaire (PRTEE) is a specific questionnaire available for assessing the health status of patients with lateral epicondylitis.
Numeric Pain Rating Scale (NPRS) | Baseline
  The Numerical Rating Scale (NPRS-11) is an 11-point scale for self-report of pain. It is the most commonly used unidimensional pain scale. The respondent selects a whole number (integers 0-10) that best reflects the intensity (or other quality if requested of his/her pain.
Numeric Pain Rating Scale (NPRS) | 8th week
  The Numerical Rating Scale (NPRS-11) is an 11-point scale for self-report of pain. It is the most commonly used unidimensional pain scale. The respondent selects a whole number (integers 0-10) that best reflects the intensity (or other quality if requested of his/her pain.
Numeric Pain Rating Scale (NPRS) | 16th week
  The Numerical Rating Scale (NPRS-11) is an 11-point scale for self-report of pain. It is the most commonly used unidimensional pain scale. The respondent selects a whole number (integers 0-10) that best reflects the intensity (or other quality if requested of his/her pain.
Numeric Pain Rating Scale (NPRS) | 6th month
  The Numerical Rating Scale (NPRS-11) is an 11-point scale for self-report of pain. It is the most commonly used unidimensional pain scale. The respondent selects a whole number (integers 0-10) that best reflects the intensity (or other quality if requested of his/her pain.

SECONDARY OUTCOMES:
Pain Pressure Threshold (PPT) | Baseline
  PPT measurement will be made using an algometer. It will be evaluated with an digital algometer over the lateral epicondyle in both upper extremities.
Pain Pressure Threshold (PPT) | 8th week
  PPT measurement will be made using an algometer. It will be evaluated with an digital algometer over the lateral epicondyle in both upper extremities.
Pain Pressure Threshold (PPT) | 16th week
  PPT measurement will be made using an algometer. It will be evaluated with an digital algometer over the lateral epicondyle in both upper extremities.
Pain Pressure Threshold (PPT) | 6th month
  PPT measurement will be made using an algometer. It will be evaluated with an digital algometer over the lateral epicondyle in both upper extremities.
Hand Grip Strength | Baseline
  Handgrip strength (HGS) is a simple and reliable measurement of maximum voluntary muscle strength. It is an important tool for diagnosing sarcopenia and is widely used as a single indicator to represent overall muscle strength. To assess grip strength, the Jamar dynamometer will be used which is recommended by the American Society for Surgery of the Hand and the American Society of Hand Therapists.
Hand Grip Strength | 8th week
  Handgrip strength (HGS) is a simple and reliable measurement of maximum voluntary muscle strength. It is an important tool for diagnosing sarcopenia and is widely used as a single indicator to represent overall muscle strength. To assess grip strength, the Jamar dynamometer will be used which is recommended by the American Society for Surgery of the Hand and the American Society of Hand Therapists.
Hand Grip Strength | 16th week
  Handgrip strength (HGS) is a simple and reliable measurement of maximum voluntary muscle strength. It is an important tool for diagnosing sarcopenia and is widely used as a single indicator to represent overall muscle strength. To assess grip strength, the Jamar dynamometer will be used which is recommended by the American Society for Surgery of the Hand and the American Society of Hand Therapists.
Hand Grip Strength | 6th month
  Handgrip strength (HGS) is a simple and reliable measurement of maximum voluntary muscle strength. It is an important tool for diagnosing sarcopenia and is widely used as a single indicator to represent overall muscle strength. To assess grip strength, the Jamar dynamometer will be used which is recommended by the American Society for Surgery of the Hand and the American Society of Hand Therapists.
Pain-free Hand Grip Strength | Baseline
  Pain-free grip strength is an important outcome measure in lateral elbow tendinopathy (LET). To assess pain-free grip strength, the Jamar dynamometer will be used which is recommended by the American Society for Surgery of the Hand and the American Society of Hand Therapists.
Pain-free Hand Grip Strength | 8th week
  Pain-free grip strength is an important outcome measure in lateral elbow tendinopathy (LET). To assess pain-free grip strength, the Jamar dynamometer will be used which is recommended by the American Society for Surgery of the Hand and the American Society of Hand Therapists.
Pain-free Hand Grip Strength | 16th week
  Pain-free grip strength is an important outcome measure in lateral elbow tendinopathy (LET). To assess pain-free grip strength, the Jamar dynamometer will be used which is recommended by the American Society for Surgery of the Hand and the American Society of Hand Therapists.
Pain-free Hand Grip Strength | 6th month
  Pain-free grip strength is an important outcome measure in lateral elbow tendinopathy (LET). To assess pain-free grip strength, the Jamar dynamometer will be used which is recommended by the American Society for Surgery of the Hand and the American Society of Hand Therapists.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No